CLINICAL TRIAL: NCT05084001
Title: Effectiveness of Silver Diamine Fluoride in Preventing Occlusal Caries in Primary Teeth of Preschool Children: a 30-month Randomized Clinical Trial
Brief Title: Silver Diamine Fluoride in Preventing Occlusal Caries in Primary Teeth
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UW20-028
Record Dates: First submitted 2021-06-08; First posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-06

CONDITIONS: Dental Caries in Children
MeSH Terms: interventions — silver diamine fluoride; Bifluorid 12

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 38% SDF (Saforide, Toyo Seiyaku Kasei Co. Ltd., Japan) (Experimental): application of silver diamine fluoride solution on occlusal surface of primary molars
  Interventions: Drug: silver diamine fluoride
- 5% NaF varnish (Duraphat, Colgate Palmolive, USA) (Active Comparator): application of sodium fluoride varnish on occlusal surface of primary molars
  Interventions: Drug: sodium fluoride varnish
- Tonic water (Placebo Comparator): application of tonic water on occlusal surface of primary molars
  Interventions: Other: tonic water

INTERVENTIONS:
Drug: silver diamine fluoride — topical application of the agent on tooth surface
  Arms: 38% SDF (Saforide, Toyo Seiyaku Kasei Co. Ltd., Japan)
Drug: sodium fluoride varnish — topical application of the agent on tooth surface
  Arms: 5% NaF varnish (Duraphat, Colgate Palmolive, USA)
Other: tonic water — topical application of tonic water on tooth surface
  Arms: Tonic water

SUMMARY:
In Hong Kong, approximately half of the kindergarten children have dental caries (tooth decay) and the majority (>90%) of the decayed teeth were left untreated. There is a need to generate clinical evidence for designing an effective dental caries prevention programme for preschool children in Hong Kong. The objective of this study is to compare the effectiveness of 38% silver diamine fluoride (SDF), 5% sodium fluoride (NaF) varnish and placebo control in preventing dentine cavitated caries in primary molars in preschool children when applied semi-annually over 30 months. Around 770 preschool children attending Grade 1 in selected kindergartens will be invited to participate in this clinical trial. Only generally healthy children with written parental consent will be included. At baseline, clinical examination will be conducted in the kindergarten to assess the tooth and oral hygiene status of the included children. After the baseline examination, the children will be randomly assigned to one of the following three study groups and the occlusal (biting) surfaces of their primary molars will receive the corresponding interventions: Group A - semi-annual topical application of 38% SDF; Group B - semi-annual application of 5% NaF varnish; and Group C - semi-annual application of placebo control with tonic water. Clinical examination of the study teeth in the children will be conducted every 6 months after the baseline to assess the outcome of the intervention. The primary outcome is whether cavitated dentine caries lesion is found in the treated occlusal tooth surface. The null hypothesis tested is that there is no difference in the effectiveness of semi-annual application of 38% SDF and that of 5% NaF varnish versus placebo control in preventing dentin occlusal caries in primary molars of preschool children. The results of the proposed study will provide evidence to strengthen or refute the recommendation regarding the use of SDF for preventing occlusal caries in primary molars. The study findings will be valuable for guiding decision-making among dental practitioners and health policymakers on whether SDF should be complemented in a school-based caries prevention program.

ELIGIBILITY:
Inclusion Criteria:

1. be healthy
2. have at least one caries-free (no cavitation) primary molar

Exclusion Criteria:

1. are uncooperative or refuse examination
2. have major systemic disease
3. present with either acute pain or infections or have gingival ulceration or stomatitis
4. have known sensitivity to fluoride, silver or other heavy-metal ions
5. are currently involved in any other research that may impact on the present study

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 769 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
dental caries increment in dmfs index | 30 months
  development of decay into dentine to form cavity

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duangthip D, He S, Gao SS, Chu CH, Lo ECM. Effectiveness of Silver Diamine Fluoride for Preventing Occlusal Caries in the Primary Teeth of Preschool Children: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2022 May 23;11(5):e35145. doi: 10.2196/35145. PMID 35604758